CLINICAL TRIAL: NCT00984659
Title: Validation of a New Shortness of Breath With Daily Activities Questionnaire in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 112989
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Results first posted 2012-03-15 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary Disease, Chronic Obstructive; Dyspnea
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Fluticasone; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- FSC (Experimental): Fluticasone propionate/salmeterol combination product 250/50mcg DISKUS twice a day
  Interventions: Drug: Fluticasone propionate/salmeterol combination product
- SAL (Experimental): Salmeterol 50mcg DISKUS twice a day
  Interventions: Drug: Salmeterol
- Placebo (Placebo Comparator): Placebo DISKUS twice a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluticasone propionate/salmeterol combination product — Fluticasone propionate/salmeterol combination product 250/50mcg DISKUS twice a day for 8 weeks
  Arms: FSC
Drug: Salmeterol — Salmeterol 50mcg DISKUS twice a day for 8 weeks
  Arms: SAL
Drug: Placebo — Placebo DISKUS twice a day for 8 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate a new questionnaire to capture the patient experience of COPD. The information collected will be used to validate the Shortness of Breath with Daily Activities Questionnaire.

DETAILED DESCRIPTION:
Dyspnea, referred to by patients as "shortness of breath" or "breathlessness," is frequently associated with decreases in functional status, quality of life, and disabilities. Currently available questionnaires do not specifically address the shortness of breath component of COPD. The development of a patient reported outcome questionnaire that will specifically assess Shortness of Breath with Daily Activities (SOBDA) in patients with COPD is needed.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 40 years of age
* Established clinical history of COPD by ATS/ERS definition
* Former or current smoker > 10 pack years
* Evidence of dyspnea

Exclusion Criteria:

* Has a respiratory disorder other than COPD
* Cancer not in complete clinical remission
* Clinically significant cardiovascular, neurological, psychiatric, renal, gastro-intestinal, immunological, endocrine, or hematological abnormalities that are uncontrolled

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2009-10-29; Primary Completion 2010-07-01 (Actual); Study Completion 2010-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (38):
- United States (38):
  - GSK Investigational Site, Jasper, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Wheat Ridge, Colorado
  - GSK Investigational Site, Stamford, Connecticut
  - GSK Investigational Site, Tamarac, Florida
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Lawrenceville, Georgia
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Madisonville, Kentucky
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Summit, New Jersey
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Elizabeth City, North Carolina
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Lake Oswego, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Chester, South Carolina
  - GSK Investigational Site, Clinton, South Carolina
  - GSK Investigational Site, Easley, South Carolina
  - GSK Investigational Site, Gaffney, South Carolina
  - GSK Investigational Site, Greenwood, South Carolina
  - GSK Investigational Site, Seneca, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Johnson City, Tennessee
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, New Braunfels, Texas
  - GSK Investigational Site, Abingdon, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Watkins ML, Wilcox TK, Tabberer M, Brooks JM, Donohue JF, Anzueto A, Chen WH, Crim C. Shortness of Breath with Daily Activities questionnaire: validation and responder thresholds in patients with chronic obstructive pulmonary disease. BMJ Open. 2013 Oct 22;3(10):e003048. doi: 10.1136/bmjopen-2013-003048. PMID 24154513
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 112989 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112989 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112989 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112989 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112989 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112989 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112989 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The number of participants "enrolled" in the Protocol reflects the number of participants starting treatment in the Double-blind Treatment Period.
Pre-assignment Details: After Screening (Visit 1), the study commenced with a 2-week Run-in Period, during which participants were permitted to use albuterol and/or ipratropium as rescue medication. Eligible participants at Visit 2 were randomized to receive one of three treatments in the 6-week Double-blind Treatment Period.
Groups:
- Albuterol and/or Ipratropium: Run-in Period: Participants were permitted to use albuterol and/or ipratropium as rescue medication during the 2-week Run-in Period
- Placebo: Double-blind Treatment Period: Matching placebo via DISKUS, administered as one inhalation twice daily (BID) during the 6-week Double-blind Treatment Period
- SAL 50 mcg: Double-blind Treatment Period: Salmeterol xinafoate (SAL) 50 micrograms (mcg) per inhalation via DISKUS, administered as one inhalation BID during the 6-week Double-blind Treatment Period
- FSC 250/50 mcg: Double-blind Treatment Period: Fluticasone propionate and salmeterol xinafoate fixed dose combination product (FSC) 250/50 mcg per inhalation via DISKUS, administered as one inhalation BID during the 6-week Double-blind Treatment Period
Period: 2-week Run-in Period
Arm/Group | Albuterol and/or Ipratropium: Run-in Period | Placebo: Double-blind Treatment Period | SAL 50 mcg: Double-blind Treatment Period | FSC 250/50 mcg: Double-blind Treatment Period
Started | 418 | 0 | 0 | 0
Completed | 366 | 0 | 0 | 0
Not Completed | 52 | 0 | 0 | 0
Not completed — Adverse Event | 8 | 0 | 0 | 0
Not completed — Protocol Violation | 5 | 0 | 0 | 0
Not completed — Study Closed/Terminated | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 3 | 0 | 0 | 0
Not completed — Physician Decision | 10 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 10 | 0 | 0 | 0
Not completed — Did Not Meet Continuation Criteria | 14 | 0 | 0 | 0
Period: 6-week Double-blind Treatment Period
Arm/Group | Albuterol and/or Ipratropium: Run-in Period | Placebo: Double-blind Treatment Period | SAL 50 mcg: Double-blind Treatment Period | FSC 250/50 mcg: Double-blind Treatment Period
Started | 0 | 75 | 152 | 139
Completed | 0 | 69 | 141 | 126
Not Completed | 0 | 6 | 11 | 13
Not completed — Adverse Event | 0 | 3 | 3 | 7
Not completed — Lack of Efficacy | 0 | 2 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 4
Not completed — Study Closed/Terminated | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 7 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Matching placebo via DISKUS, administered as one inhalation twice daily (BID)
- SAL 50 mcg: Salmeterol xinafoate (SAL) 50 micrograms (mcg) per inhalation via DISKUS, administered as one inhalation BID
- FSC 250/50 mcg: Fluticasone propionate and salmeterol xinafoate fixed dose combination product (FSC) 250/50 mcg per inhalation via DISKUS, administered as one inhalation BID
- Albuterol and/or Ipratropium: Run-in Failure: Participants who entered the 2-week Run-in Period, during which they were permitted to use albuterol and/or ipratropium as rescue medication, but then failed to be randomized, or were randomized but did not receive a dose of study medication
- Total: Total of all reporting groups
Arm/Group | Placebo | SAL 50 mcg | FSC 250/50 mcg | Albuterol and/or Ipratropium: Run-in Failure | Total
Number analyzed (Participants) | 75 | 152 | 139 | 52 | 418
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.8 (9.82) | 60.1 (9.58) | 60.2 (9.45) | 63.8 (9.61) | 61.1 (9.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 63 | 60 | 27 | 179
  Male | 46 | 89 | 79 | 25 | 239
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 9 | 12 | 12 | 8 | 41
  Asian | 1 | 0 | 0 | 0 | 1
  White | 65 | 140 | 127 | 44 | 376

OUTCOME MEASURES:

1. Primary Outcome: Internal Consistency (IC) of the Shortness of Breath With Daily Activities (SOBDA) Questionnaire in Participants With Chronic Obstructive Pulmonary Disease (COPD) Assessed as Cronbach's Alpha Value
Description: Cronbach's alpha (CA) is a measure of the IC of the 13-item SOBDA questionnaire (completed via electronic diary by a sample of participants). It is the ratio of the variance (var.) of the sum of the individual scores and the var. of the total score. The var. of the sum of a group of independent variables is the sum of their var.; thus, if the variables are positively correlated, the var. of the sum will be increased. If the items making up the score are identical and so perfectly correlated, CA=1. If the items are independent, CA=0. Higher scores indicate a more reliable (precise) instrument.
Time Frame: Day 1 of the 2-week Run-in Period
Population: Run-in Population: all participants who completed Visit 2 (Day 1 of Treatment Period), including those who were not randomized, were randomized but did not receive a dose of study medication, and those who were randomized and received study medication. Participants with a score for each SOBDA item on Day 1 of the 2-week Run-in Period were analyzed.
Measure: Number; unit: ratio of variance
Groups:
- All Participants: 2-week Run-in Period: All participants in the 2-week Run-in Period. Participants were permitted to use albuterol and/or ipratropium as rescue medication during this period.
Arm/Group | All Participants: 2-week Run-in Period
Number analyzed (Participants) | 344
ratio of variance | 0.892

2. Primary Outcome: Test-retest Reliability (T-RR) of SOBDA Scores Measured as the Difference in the SOBDA Weekly Score Between Week 1 and Week 2 of the 2-week Run-in Period
Description: T-RR=stability during repeat measures over time in a stable population. SOBDA score was determined by the 13-item (it.) scoring algorithm, assigning a weekly mean score of 1-4 (higher scores=more severe breathlessness with daily activities) based on the mean of 7 days of data (or >=4 days). Daily total score is computed from the mean of the participant's (par.) scores on the 13 it. (>=7 it. must have non-missing responses). Only scores of stable par. (indicating no change [score=3] on the par.-completed Patient Global Assessment of Change [PGAC]; 1 [ much worse] to 5 [much better]) were used.
Time Frame: Week 1 and Week 2 of the 2-week Run-in Period
Population: Run-in Population. Data from participants with weekly SOBDA scores at Week 1 and Week 2 of the 2-week Run-in Period and reporting no change on the second weekly PGAC were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | All Participants: 2-week Run-in Period
Number analyzed (Participants) | 152
scores on a scale | 0.01 (0.244)
Statistical Analysis 1: Comparison: All Participants: 2-week Run-in Period; Test type: Superiority or Other; p = 0.713, t-test, 2 sided; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.03 to 0.05]

3. Primary Outcome: Convergent Validity for the SOBDA Questionnaire Measured as Correlations of the Baseline SOBDA Score With Participant-completed Modified Medical Research Council (mMRC) and Physician-completed mMRC Scores at Visit 2
Description: Convergent validity is defined as the ability of the SOBDA questionnaire to measure required information and was assessed by examining the relationship between the SOBDA score and the participant/physician-completed mMRC Dyspnea Scale assessments. The physician/participant rated the degree of the participant's dyspnea (trouble breathing) on the 5-point mMRC scale (0, none; 4, very severe). Spearman's rank correlation coefficient assesses if the relationship between two variables is monotone. A correlation of +1 or -1 will occur if one variable is a perfect monotone of the other.
Time Frame: Baseline (last week of the 2-week Run-in Period) and pre-treatment on Visit 2 (Day 1 of the 6-week Treatment Period)
Population: Run-in Population. Participants with a SOBDA Baseline score and the indicated assessment at Visit 2 were analyzed. One participant who rated their own trouble breathing had missing data for the physician assessment.
Measure: Number; unit: Spearman rank correlation coefficient
Arm/Group | All Participants: 2-week Run-in Period
Number analyzed (Participants) | 340
Spearman rank correlation coefficient
  Physician-completed mMRC, n=339 | 0.24
  Participant-completed mMRC, n=340 | 0.29

4. Primary Outcome: Convergent Validity for the SOBDA Questionnaire Measured as the Correlation of the Baseline SOBDA Score With the Clinician Global Assessment of Dyspnea Severity (CGI-S) Score at Visit 2
Description: Convergent validity is defined as the ability of the SOBDA questionnaire to measure the required information and was assessed by examining the relationship between the SOBDA score with the CGI-S score. Spearman's rank correlation coefficient assesses if the relationship between two variables is monotone. A correlation of +1 or -1 will occur if one variable is a perfect monotone of the other. Clinicians were asked to assess the severity of the participant's dyspnea on the CGI-S scale. This was evaluated on a 1-4 Likert scale: 1 (mild) to 4 (very severe).
Time Frame: Baseline (last week of the 2-week Run-in Period) and pre-treatment on Visit 2 (Day 1 of the 6-week Treatment Period)
Population: Run-in Population. Participants with a SOBDA Baseline score and the indicated assessment at Visit 2 were analyzed.
Measure: Number; unit: Spearman rank correlation coefficient
Arm/Group | All Participants: 2-week Run-in Period
Number analyzed (Participants) | 338
Spearman rank correlation coefficient | 0.24

5. Primary Outcome: Convergent Validity (CV) for the SOBDA Questionnaire Measured as the Correlation of the Baseline SOBDA Score With the Chronic Respiratory Disease Questionnaire-Self-Administered Standardized (CRQ-SAS) Dyspnea Domain Score at Visit 2
Description: Convergent validity is defined as the ability of the SOBDA questionnaire to measure required information and was assessed by examining the relationship between the SOBDA score and the CRQ-SAS dyspnea domain score. Pearson's correlation coefficient is a measure of the linear dependence between 2 variables. A correlation of +1 or -1 will occur if the data from the 2 variables lie exactly on a line. The CRQ is a 20-item instrument measuring 4 domains (each measured on a scale of 1 [maximum impairment] to 7 [no impairment]) of functioning: mastery, fatigue, emotional function, and dyspnea.
Time Frame: Baseline (last week of the 2-week Run-in Period) and pre-treatment on Visit 2 (Day 1 of the 6-week Treatment Period)
Population: Run-in Population. Participants with a SOBDA Baseline score and the indicated assessment at Visit 2 were analyzed.
Measure: Number; unit: Pearson's correlation coefficient
Arm/Group | All Participants: 2-week Run-in Period
Number analyzed (Participants) | 340
Pearson's correlation coefficient | -0.68

6. Primary Outcome: Known Group Validity for the SOBDA Questionnaire Measured as the Comparison of the Baseline SOBDA Score in the Indicated Categories of the Physician-completed (PyC) mMRC Score at Visit 2
Description: SOBDA known group validity refers to the extent to which scores from the SOBDA questionnaire should differentiate participants with varying levels of dyspnea severity. It was assessed by comparing summary measures for the SOBDA score for each indicated level (0, 1, 2, 3, and 4) of the PyC mMRC. The physician rated the degree of the participant's dyspnea on the 5-point mMRC scale: 0 (none) to 4 (very severe). Known group validity was confirmed if the SOBDA score increased with increasing values of PyC mMRC, both indicating increased levels of breathlessness.
Time Frame: Baseline (last week of the 2-week Run-in Period) and pre-treatment on Visit 2 (Day 1 of the 6-week Treatment Period)
Population: Run-in Population. Participants with a SOBDA Baseline score and the Physician-completed mMRC score at Visit 2 were analyzed.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | All Participants: 2-week Run-in Period
Number analyzed (Participants) | 339
scores on a scale
  PyC mMRC: 0 to 1, n=12 | 1.78 (0.196)
  PyC mMRC: 2, n=200 | 2.08 (0.048)
  PyC mMRC: 3, n=117 | 2.28 (0.063)
  PyC mMRC: 4, n=10 | 2.73 (0.216)
Statistical Analysis 1: Comparison: All Participants: 2-week Run-in Period; Test type: Superiority or Other; p < 0.001, ANCOVA — Analysis of covariance (ANCOVA) adjusted for age, gender, and percent predicted Forced Expiratory volume in one second (FEV1) at Screening

7. Primary Outcome: Known Group Validity for the SOBDA Questionnaire Measured as the Comparison of the Baseline SOBDA Score in the Indicated Categories of the Participant-completed (ParC) mMRC Score at Visit 2
Description: SOBDA known group validity refers to the extent to which scores from the SOBDA questionnaire should differentiate participants with varying levels of dyspnea severity. It was assessed by comparing summary measures for the SOBDA score for each indicated level (0, 1, 2, 3, and 4) of the ParC mMRC. The participant rated the degree of his/her dyspnea on the 5-point mMRC scale: 0 (none) to 4 (very severe). Known group validity was confirmed if the SOBDA score increased with increasing values of ParC mMRC, both indicating increased levels of breathlessness.
Time Frame: Baseline (last week of the 2-week Run-in Period) and pre-treatment on Visit 2 (Day 1 of the 6-week Treatment Period)
Population: Run-in Population. Participants with a SOBDA Baseline score and the Participant-completed mMRC score at Visit 2 were analyzed.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | All Participants: 2-week Run-in Period
Number analyzed (Participants) | 340
scores on a scale
  ParC mMRC: 0, n=12 | 1.92 (0.192)
  ParC mMRC: 1, n=103 | 1.94 (0.066)
  ParC mMRC: 2, n=138 | 2.20 (0.056)
  ParC mMRC: 3, n=65 | 2.26 (0.083)
  ParC mMRC: 4, n=22 | 2.73 (0.142)
Statistical Analysis 1: Comparison: All Participants: 2-week Run-in Period; Test type: Superiority or Other; p < 0.001, ANCOVA — ANCOVA adjusted for age, gender, and percent predicted FEV1 at Screening

8. Primary Outcome: Known Group Validity (KGV) for the SOBDA Questionnaire Measured as the Comparison of the Baseline SOBDA Score in the Indicated Categories of CGI-S Scores at Visit 2
Description: SOBDA KGV refers to the extent to which scores from the SOBDA questionnaire should differentiate participants with varying levels of dyspnea severity. It was assessed by comparing summary measures for the SOBDA score for each indicated level (0, 1, 2, 3, and 4) of the CGI-S score. Clinicians were asked to assess the severity of the participant's dyspnea on the CGI-S scale. This was evaluated on a 1-4 Likert scale: 1 (mild) to 4 (very severe). KGV was confirmed if the SOBDA score increased with increasing values of CGI-S, both indicating increased levels of breathlessness.
Time Frame: Baseline (last week of the 2-week Run-in Period) and pre-treatement on Visit 2 (Day 1 of the 6-week Treatment Period)
Population: Run-in Population. Participants with a SOBDA Baseline score and the CGI-S score at Visit 2 were analyzed.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | All Participants: 2-week Run-in Period
Number analyzed (Participants) | 338
scores on a scale
  CGI-S: 1, n=19 | 1.87 (0.156)
  CGI-S: 2, n=236 | 2.11 (0.045)
  CGI-S: 3, n=78 | 2.33 (0.080)
  CGI-S: 4, n=5 | 2.72 (0.305)
Statistical Analysis 1: Comparison: All Participants: 2-week Run-in Period; Test type: Superiority or Other; p = 0.008, ANCOVA — ANCOVA adjusted for age, gender, and percent predicted FEV1 at Screening

9. Primary Outcome: Participants (Par.) Classified as Responders/Non-responders According to the Patient Global Assessment of Change (PGAC) Response at Days 8, 15, 22, 29, 36, and 43 and at Visit 3/Premature Discontinuation (PD) (the End of the 6-week Treatment Period or PD)
Description: The PGAC is par. completed on a 1-5 scale: 1, much worse; 2, worse; 3, no change; 4, better; 5, much better. Responders were defined as par. with a rating of "better" or "much better" (score of 4 or 5) on the PGAC at the relevant week; non-responders were defined as par. with a response of "much worse," "worse," or "no change" on the PGAC. As pre-specified in the study protocol, results are presented independent of treatment allocation . The study objectives were to assess the measurement properties and validity of the SOBDA questionnaire independent of specific treatment effect.
Time Frame: Days 8, 15, 22, 29, 36, and 43 and Visit 3/PD (end of 6-week Treatment Period or earlier up to Week 8)
Population: Modified Intent-to-Treat (MITT) Population: all participants randomized to treatment who received at least one dose of study medication. Analyses were conducted on data available for each specified time point.
Measure: Number; unit: participants
Groups:
- MITT Population: 6-Week Treatment Period: Participants randomized to receive FSC 250/50 mcg BID, SAL 50 mcg BID, or placebo BID for the 6-week Treatment Period comprising the MITT Population
Arm/Group | MITT Population: 6-Week Treatment Period
Number analyzed (Participants) | 303
participants
  Responders, Day 8 (Baseline to Week 1), n=293 | 105
  Non-responders, Day 8 (Baseline to Week 1), n=293 | 188
  Responders, Day 15 (Week 1 to Week 2), n=303 | 91
  Non-responders, Day 15 (Week 1 to Week 2), n=303 | 212
  Responders, Day 22 (Week 2 to Week 3), n=299 | 83
  Non-responders, Day 22 (Week 2 to Week 3), n=299 | 216
  Responders, Day 29 (Week 3 to Week 4), n=285 | 62
  Non-responders, Day 29 (Week 3 to Week 4), n=285 | 223
  Responders, Day 36 (Week 4 to Week 5), n=277 | 77
  Non-responders, Day 36 (Week 4 to Week 5), n=277 | 200
  Responders, Day 43 (Week 5 to Week 6), n=119 | 31
  Non-responders, Day 43 (Week 5 to Week 6), n=119 | 88
  Responders, Last Treatment Week, n=151 | 45
  Non-responders, Visit 3/PD, n=151 | 106

10. Primary Outcome: Change From the Previous Week to the Current Week's SOBDA Score by Participant-completed PGAC Response at Days 8, 15, 22, 29, 36, and 43 and at Visit 3/PD (End of the 6-week Treatment Period or PD)
Description: Responsiveness reflects the ability of the SOBDA questionnaire to detect change under conditions of known change. Responders (Rs)=participants (par.) with a rating of "better"/"much better" (score of 4/5) on the PGAC (range; 1 [much worse] to 5 [much better]) at the relevant week; NRs=par. with a response of "much worse," "worse," or "no change" (score of 3). Mean difference between Rs and NRs in the change from the previous week to the current week's SOBDA score was calculated. For Visit 3/PD, the change from Baseline to the last treatment week's SOBDA score for Rs and NRs was calculated.
Time Frame: Baseline; Days 8, 15, 22, 29, 36, and 43 and Visit 3/PD (end of 6-week Treatment Period or earlier up to Week 8)
Population: MITT Population. Analyses were conducted on data available for each specified time point. As pre-specified in the study protocol, results are presented independent of treatment allocation. The study objectives were to assess the measurement properties and validity of the SOBDA questionnaire independent of specific treatment effect.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | MITT Population: 6-Week Treatment Period
Number analyzed (Participants) | 223
scores on a scale
  Baseline to Day 8, responders, n=105 | -0.26 (0.324)
  Baseline to Day 8, non-responders, n=188 | -0.01 (0.254)
  Day 8 to Day 15, responders, n=91 | -0.10 (0.280)
  Day 8 to Day 15, non-responders, n=212 | 0.01 (0.222)
  Day 15 to Day 22, responders, n=83 | -0.08 (0.223)
  Day 15 to Day 22, non-responders, n=216 | 0.02 (0.183)
  Day 22 to Day 29, responders, n=62 | -0.09 (0.198)
  Day 22 to Day 29, non-responders, n=223 | 0.01 (0.193)
  Day 29 to Day 36, responders, n=77 | -0.07 (0.245)
  Day 29 to Day 36, non-responders, n=200 | 0.03 (0.169)
  Day 36 to Day 43, responders, n=31 | -0.04 (0.167)
  Day 36 to Day 43, non-responders, n=88 | 0.02 (0.240)
  Baseline to Visit 3/PD, responders, n=45 | -0.21 (0.497)
  Baseline to Visit 3/PD, non-responders, n=106 | -0.14 (0.423)
Statistical Analysis 1: Comparison: MITT Population: 6-Week Treatment Period; Test type: Superiority or Other; p < 0.001, ANCOVA — ANCOVA adjusted for age, gender, and SOBDA Baseline score; difference between responders and non-responders during Week prior to Day 8; Mean Difference (Final Values) = 0.24, 95% CI [0.18 to 0.31]
Statistical Analysis 2: Comparison: MITT Population: 6-Week Treatment Period; Test type: Superiority or Other; p < 0.001, ANCOVA — ANCOVA adjusted for age, gender, and SOBDA Baseline score; difference between responders and non-responders during Week prior to Day 15; Median Difference (Final Values) = 0.12, 95% CI [0.06 to 0.19]
Statistical Analysis 3: Comparison: MITT Population: 6-Week Treatment Period; Test type: Superiority or Other; p < 0.001, ANCOVA — ANCOVA adjusted for age, gender, and SOBDA Baseline score; difference between responders and non-responders during Week prior to Day 22; Mean Difference (Final Values) = 0.11, 95% CI [0.06 to 0.16]
Statistical Analysis 4: Comparison: MITT Population: 6-Week Treatment Period; Test type: Superiority or Other; p < 0.001, ANCOVA — ANCOVA adjusted for age, gender, and SOBDA Baseline score; difference between responders and non-responders during Week prior to Day 29; Mean Difference (Final Values) = 0.11, 95% CI [0.06 to 0.17]
Statistical Analysis 5: Comparison: MITT Population: 6-Week Treatment Period; Test type: Superiority or Other; p < 0.001, ANCOVA — ANCOVA adjusted for age, gender, and SOBDA Baseline score; difference between responders and non-responders during Week prior to Day 36; Mean Difference (Final Values) = 0.13, 95% CI [0.08 to 0.18]
Statistical Analysis 6: Comparison: MITT Population: 6-Week Treatment Period; Test type: Superiority or Other; p = 0.180, ANCOVA — ANCOVA adjusted for age, gender, and SOBDA Baseline score; difference between responders and non-responders during Week prior to Day 43; Mean Difference (Final Values) = 0.06, 95% CI [-0.03 to 0.15]
Statistical Analysis 7: Comparison: MITT Population: 6-Week Treatment Period; Test type: Superiority or Other; p = 0.307, ANCOVA — ANCOVA adjusted for age, gender, and SOBDA Baseline score; difference between responders and non-responders during Week prior to Visit 3/PD; Mean Difference (Final Values) = 0.08, 95% CI [-0.07 to 0.23]

11. Primary Outcome: Number of Participants Classified as Responders and Non-responders by Clinician Global Impression of Change Question (CGI-C) Response at Visit 3/PD
Description: Clinicians were asked to provide their clinical impression regarding change in the participant's shortness of breath by CGI-C. This was evaluated on a 1-5 Likert scale: 1 (much worse) to 5 (much better), with 3 being no change. A CGI-C responder was defined as a participant who had a response of "better" (4) or "much better" (5), and a non-responder was defined as a participant who had a response of "much worse" (1), "worse" (2), or "no change" (3).
Time Frame: Visit 3/PD (end of 6-week Treatment Period or earlier up to Week 8)
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | MITT Population: 6-Week Treatment Period
Number analyzed (Participants) | 301
participants
  Responders | 120
  Non-responders | 181

12. Primary Outcome: Number of Participants Classified as Responders and Non-responders by CRQ-SAS Dyspnea Domain Response at Visit 3/PD
Description: A CRQ-SAS dyspnea domain responder was defined as a participant who had a score increase of 0.5 units or more for the dyspnea domain of the CRQ-SAS between Visit 2 and Visit 3/Premature Discontinuation. A non-responder was defined as a participant who had a decrease in the score, or an increase of less than 0.5 units.
Time Frame: Visit 3/PD (end of 6-week Treatment Period or earlier up to Week 8)
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | MITT Population: 6-Week Treatment Period
Number analyzed (Participants) | 301
participants
  Responders | 117
  Non-responders | 184

13. Primary Outcome: Number of Participants Classified as Responders and Non-responders by Physician-completed and Participant-completed mMRC Response at Visit 3/PD
Description: A Physician-completed and Participant-completed mMRC responder was defined as a participant who had a score decrease of one unit or more between Visit 2 and Visit 3/Premature Discontinuation. A non-responder was defined as a participant who had the same score or an increase in score.
Time Frame: Visit 3/PD (end of 6-week Treatment Period or earlier up to Week 8)
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | MITT Population: 6-Week Treatment Period
Number analyzed (Participants) | 301
participants
  Physician-completed mMRC responders | 91
  Physician-completed mMRC non-responders | 210
  Participant-completed mMRC responders | 92
  Participant-completed mMRC non-responders | 209

14. Primary Outcome: Change From Baseline to Last Treatment Week in the SOBDA Score by CGI-C Responses at Visit 3/PD
Description: The responsiveness of the SOBDA questionnaire was assessed by comparing score changes between responders and non-responders. The CGI-C is clinician completed on a 1 to 5 scale: 1, much worse; 2, worse; 3, no change; 4, better; 5, much better. Changes in mean SOBDA scores during the last week of treatment in responders and non-responders using definitions based on the CGI-C conducted at Visit 3/Premature Discontinuation were assessed.
Time Frame: Baseline (2-week Run-in Period) and Week Prior to Visit 3/PD (end of 6-week Treatment Period or earlier up to Week 8)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | MITT Population: 6-Week Treatment Period
Number analyzed (Participants) | 301
scores on a scale
  Responders, n=120 | -0.25 (0.484)
  Non-responders, n=181 | -0.03 (0.413)
Statistical Analysis 1: Comparison: MITT Population: 6-Week Treatment Period; Test type: Superiority or Other; p < 0.001, ANCOVA — ANCOVA adjusted for age, gender, and SOBDA Baseline score; comparision of mean SOBDA score for CGI-C responders and non-responders; Mean Difference (Final Values) = 0.24, 95% CI [0.14 to 0.34]

15. Primary Outcome: Change From Baseline to Last Treatment Week in the SOBDA Score by CRQ-SAS Dyspnea Domain (DD) Responses at Visit 3/PD
Description: The responsiveness of the SOBDA questionnaire was assessed by comparing score changes of responders (Rs) versus non-responders (NRs). The CRQ-SAS DD includes 5 questions (q.) scored 1 (maximum impairment) to 7 (no impairment). Individual q. were equally weighted, and domain scores (DSs) (range=1-7) were calculated as the mean across the non-missing items within each domain (DSs were calculated although an individual item score was missing). Changes in mean SOBDA scores during the last treatment week in Rs and NRs using definitions based on the CRQ-SAS DD conducted at Visit 3/PD were assessed.
Time Frame: Baseline (2-week Run-in Period) and Week Prior to Visit 3/PD (end of 6-week Treatment Period or earlier up to Week 8)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | MITT Population: 6-Week Treatment Period
Number analyzed (Participants) | 301
Scores on a scale
  Responders, n=117 | -0.32 (0.446)
  Non-responders, n=184 | 0.01 (0.416)
Statistical Analysis 1: Comparison: MITT Population: 6-Week Treatment Period; Test type: Superiority or Other; p < 0.001, ANCOVA — ANCOVA adjusted for age, gender, and SOBDA Baseline score; comparision of mean SOBDA score for CRQ-SAS Dyspnea Domain responders and non-responders; Median Difference (Final Values) = 0.30, 95% CI 2-sided [0.21 to 0.40]

16. Primary Outcome: Change From Baseline to Last Treatment Week in the SOBDA Score by Physician-completed mMRC and Participant-completed mMRC Responses at Visit 3/PD
Description: The responsiveness of the SOBDA questionnaire was assessed by comparing score changes between responders and non-responders. The mMRC ranges from 0 (no breathlessness except with strenous exercise) to 4 (too breathless to leave the house; breathless when dressing/undressing) and is completed by the clinician or the participant as indicated. Changes in mean SOBDA scores during the last week of treatment in responders and non-responders using definitions based on the Physician-completed (Ph-C) and Participant-completed (Pa-C) mMRC conducted at Visit 3/Premature Discontinuation were assessed.
Time Frame: Baseline (2-week Run-in Period) and Week Prior to Visit 3/PD (end of 6-week Treatment Period or earlier up to Week 8)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | MITT Population: 6-Week Treatment Period
Number analyzed (Participants) | 301
Scores on a scale
  Ph-C mMRC, responders, n=91 | -0.13 (0.416)
  Ph-C mMRC, non-responders, n=210 | -0.11 (0.472)
  Pa-C mMRC, responders, n=92 | -0.18 (0.508)
  Pa-C mMRC, non-responders, n=209 | -0.09 (0.428)
Statistical Analysis 1: Comparison: MITT Population: 6-Week Treatment Period; Test type: Superiority or Other; p = 0.535, ANCOVA — ANCOVA adjusted for age, gender, and SOBDA Baseline score; comparision of mean SOBDA score for Physician-Completed mMRC responders and non-responders; Median Difference (Final Values) = 0.03, 95% CI [-0.08 to 0.15]
Statistical Analysis 2: Comparison: MITT Population: 6-Week Treatment Period; Test type: Superiority or Other; p = 0.08, ANCOVA — ANCOVA adjusted for age, gender, and SOBDA Baseline score; comparison of mean SOBDA score for Participant-Completed mMRC responders and non-responders; Median Difference (Final Values) = 0.08, 95% CI [-0.02 to 0.19]

17. Primary Outcome: SOBDA Threshold for Response Assessed as Mean Change From the Previous Week's SOBDA Score Based on a Participant-completed PGAC Score Rated of "Better"
Description: Changes from Baseline in the SOBDA score for responders (Rs) and non-responders (NRs) (using the PGAC assessment; 1 [much worse] to 5 [much better]), together with the cumulative proportions of Rs and NRs, was used to establish the threshold for defining SOBDA questionnaire Rs. The threshold of response is a score change in the SOBDA questionnaire that is demonstrated to have a perceivable benefit for the participant. The threshold of response was evaluated as the change from Baseline in the SOBDA score based on PGAC scores pre-specified as "better" or demonstrating meaningful improvement.
Time Frame: Baseline (last week of the 2-week Run-in Period) and Weeks 1, 2, 3, 4, 5, and 6 (6-week Treatment Period)
Population: MITT Population. Analyses were conducted on data available for each specified time point. As pre-specified in the study protocol, results are presented independent of treatment allocation . The study objectives were to assess the measurement properties and validity of the SOBDA questionnaire independent of specific treatment effect.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | MITT Population: 6-Week Treatment Period
Number analyzed (Participants) | 97
scores on a scale
  Baseline to Week 1, n=97 | -0.26 (0.325)
  Week 1 to Week 2, n=82 | -0.08 (0.219)
  Week 2 to Week 3, n=70 | -0.08 (0.216)
  Week 3 to Week 4, n=49 | -0.10 (0.216)
  Week 4 to Week 5, n=66 | -0.08 (0.255)
  Week 5 to Week 6, n=26 | -0.05 (0.181)

18. Primary Outcome: SOBDA Threshold for Response as Assessed by Mean Change From Baseline to the Last Treatment Week in the SOBDA Score Based on a CGI-C Response Rated as "Better"
Description: The threshold of response is a score change in the SOBDA questionnaire that is demonstrated to have a perceivable benefit for the participant. The threshold of response was evaluated as the change from Baseline in the SOBDA score based on CGI-C scores pre-specified as "better" or demonstrating meaningful improvement. The CGI-C is clinician completed on a 1 to 5 scale: 1, much worse, 2, worse; 3, no change; 4, better; 5, much better.
Time Frame: Baseline and Week Prior to Visit 3/PD (end of 6-week Treatment Period or earlier up to Week 8)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | MITT Population: 6-Week Treatment Period
Number analyzed (Participants) | 109
Scores on a scale | -0.25 (0.484)

19. Primary Outcome: SOBDA Threshold for Response as Assessed by Mean Change From Baseline to the Last Treatment Week in the SOBDA Score Based on a CRQ-SAS Dyspnea Domain (DD) Response Rated as "Better"
Description: The threshold of response (TOR) is a score change in the SOBDA questionnaire that is demonstrated to have a perceivable benefit. The TOR was evaluated as the change from Baseline in the SOBDA score based on CRQ-SAS scores pre-specified as "better" or demonstrating meaningful improvement. The CRQ-SAS DD includes 5 questions (q.) scored 1 (maximum impairment) to 7 (no impairment). Individual q. were equally weighted, and domain scores (DSs) (range=1-7) were calculated as the mean across the non-missing items within each domain (DSs were calculated although an individual item score was missing).
Time Frame: Baseline and Week Prior to Visit 3/PD (end of 6-week Treatment Period or earlier up to Week 8)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | MITT Population: 6-Week Treatment Period
Number analyzed (Participants) | 68
Scores on a scale | -0.13 (0.417)

20. Primary Outcome: SOBDA Threshold for Response Assessed as Mean Change From Baseline to Last Treatment Week in the SOBDA Score Based on Forced Expiratory Volume in One Second (FEV1) Change From Baseline of 50 Milliliters (mL) to <100 mL
Description: FEV1 response was rated as 1=No change or worse (i.e., change of <50 mL); 2=Better (i.e., change of 50 to <100 mL); 3=Much better (i.e., change of >=100 mL). The threshold of response is a score change in the SOBDA questionnaire that is demonstrated to have a perceivable benefit for the participant. The threshold of response was evaluated as the change from Baseline in the SOBDA score based on study assessment (FEV1) scores pre-specified as "better" or demonstrating meaningful improvement.
Time Frame: Baseline and Week Prior to Visit 3/PD (end of 6-week Treatment Period or earlier up to Week 8)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | MITT Population: 6-Week Treatment Period
Number analyzed (Participants) | 42
mL | -0.16 (0.492)

ADVERSE EVENTS:
Description: Safety data are presented for the Modified Intent-to-Treat (MITT) Population, comprised of all participants randomized to treatment who received at least one dose of study medication. Data summaries and analyses were based on the actual treatment received. One participant in the SAL 50 mcg arm was randomized but did not receive treatment.
Groups:
- FSC 250/50 mcg: Fluticasone propionate and salmeterol xinafoate fixed dose combination product (FSC) 250/50 mcg per inhalation via DISKUS, administered as one inhalation BID during the 6-week Double-blind Treatment Period
Arm/Group | Placebo | SAL 50 mcg | FSC 250/50 mcg
Serious Adverse Events (participants affected / at risk) | 4/75 | 5/151 | 3/139
Other Adverse Events (participants affected / at risk) | 14/75 | 34/151 | 37/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=75) | SAL 50 mcg (N=151) | FSC 250/50 mcg (N=139)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1
Impaired Gastric Emptying (Gastrointestinal disorders) | 0 | 1 | 0
Chest Pain (General disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 0 | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 1 | 0
Suicide Attempt (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=75) | SAL 50 mcg (N=151) | FSC 250/50 mcg (N=139)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Candidiasis (Infections and infestations) | 1 | 0 | 3
Nasopharyngitis (Infections and infestations) | 1 | 2 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 1
Gastroenteritis Viral (Infections and infestations) | 0 | 1 | 1
Influenza (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 2 | 0
Respiratory Tract Infection (Infections and infestations) | 2 | 0 | 0
Acute Sinusitis (Infections and infestations) | 0 | 0 | 1
Gastric Infection (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Pneumonia Klebsiella (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 6 | 5
Sinus Headache (Nervous system disorders) | 0 | 0 | 3
Carpal tunnel Syndrome (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Impaired Gastric Emptying (Gastrointestinal disorders) | 0 | 1 | 0
Lip Swelling (Gastrointestinal disorders) | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Lower Extremity Mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Chest Pain (General disorders) | 1 | 3 | 0
Adverse Drug Reaction (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0
Irritability (General disorders) | 0 | 0 | 1
Edema Peripheral (General disorders) | 1 | 0 | 0
Pain (General disorders) | 0 | 1 | 0
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Ankle Fracture (General disorders) | 0 | 0 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint Sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperlipidemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 2 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Nervousness (Psychiatric disorders) | 1 | 0 | 0
Suicide Attempt (Psychiatric disorders) | 0 | 0 | 1
Blood Pressure Increased (Investigations) | 1 | 0 | 1
Heart Rate Increased (Investigations) | 0 | 1 | 0
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Seborrhoeic Keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Periorbital Edema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 1
Vision Blurred (Eye disorders) | 0 | 0 | 1
Multiple Allergies (Immune system disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.